CLINICAL TRIAL: NCT00470834
Title: A Randomized Double-Blind Parallel Group Study Comparing Casodex (or Generic Equivalent) 50mg Plus Placebo to Casodex (or Generic Equivalent) 50mg Plus Dutasteride 3.5mg Administered for 18 Months to Men With Prostate Cancer Who Have Failed First-Line Androgen Deprivation Therapy (Assessed by Rising PSA) Followed by a Two-Year Extension Phase
Brief Title: Prostate Cancer Study In Men Who Have Failed First-Line Androgen Deprivation Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVO108943
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Results first posted 2013-11-01 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2016-11

CONDITIONS: Neoplasms, Prostate
Keywords: prostate cancer; androgen deprivation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dutasteride; bicalutamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): 50 mg bicalutamide and 3.5 mg Dutasteride (IP)
  Interventions: Drug: dutasteride; Drug: bicalutamide
- Arm 2 (Placebo Comparator): 50 mg bicalutamide and placebo
  Interventions: Drug: placebo; Drug: bicalutamide

INTERVENTIONS:
Drug: dutasteride — 0.5mg dutasteride (Investigation Product)
  Arms: Arm 1
Drug: placebo — making placebo
  Arms: Arm 2
Drug: bicalutamide — 50 mg Casodex or generic equivalent

SUMMARY:
Dutasteride inhibits the conversion of testosterone to dihydrotestosterone (DHT) the male hormone that leads to benign prostate growth. By blocking the conversion of testosterone to DHT, dutasteride could allow bicalutamide to be a more effective anti-androgen thus prolonging bicalutamide's efficacy.

ELIGIBILITY:
Inclusion criteria:

* Men ≥40 and ≤90 years of age
* Must have asymptomatic prostate cancer that has progressed during androgen deprivation therapy (rising PSA). PSA progression must have occurred after first-line treatment with GnRH analogues ( e.g. leuprolide, goserelin) or orchiectomy. PSA progression is defined by three rises in PSA each measured at least 4 weeks apart within the previous year.
* Serum PSA ≥2 and ≤20ng/ml from central laboratory. One PSA retest from central laboratory is allowed if the value is <2 or >20ng/ml; or if the PSA value is not consistent with the previous rising PSA values that determined progression while on a GnRH analogue.
* Serum Testosterone <50ng/ml from central laboratory.
* Non-metastatic prostate cancer as confirmed on prior bone scan performed within 8 weeks of screening.
* Expected survival ≥ 2 years
* ECOG Performance status 0, 1, or 2

Exclusion criteria:

* Additional hormonal therapy (excluding the current use of a GnRH analogue) within the past 6 months of:
* Estrogens (e.g. megestrol, medroxyprogesterone, cyproterone, DES)
* Drugs with antiandrogenic properties (e.g., spironolactone if >50mg/day, flutamide, bicalutamide*, ketoconazole**, progestational agents)

  *The use of an antiandrogen during GnRH analogue induction for <6 weeks is acceptable, but none within the 3 months prior to study entry.

  **The use of topical ketoconazole is permitted prior to and during the study. NOTE: Use of dietary and herbal supplements (e.g., selenium, Vitamin E, saw palmetto), excluding daily vitamins, during the study is discouraged, but not prohibited. All dietary and herbal supplement usage will be recorded in the eCRF.
* Treatment with oral glucocorticoids during the 3 months prior to randomization or expectation of their use during the study.
* Prior chemotherapy for prostate cancer. (prior prostatectomy or radiotherapy to the prostate are allowed)
* Prostate surgery including TUNA, TURP, TUIP, laser treatment, thermotherapy, balloon dilatation, prosthesis, and cryosurgical ablation within 2 months prior to enrollment.
* Current and/or previous use of the following medications:
* Finasteride (Proscar, Propecia), or Dutasteride (GI198745, AVODART) exposure within 6 months prior to study entry
* Anabolic steroids (within 6 months prior to study entry)
* Participation in any investigational or marketed drug trial within the 30 days prior to the first dose of study drug or anytime during the study period.
* Any unstable serious co-existing medical condition(s) including but not limited to myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident within 6 months prior to Screening visit; uncontrolled diabetes; or peptic ulcer disease which is uncontrolled by medical management.
* Abnormal liver function test greater than 1.5 times the upper limit of normal for alanine aminotransferase [ALT], aspartate aminotransferase [AST], alkaline phosphatase [ALP] or bilirubin.
* Serum creatinine >2.0 times the upper limit of normal.
* History of another malignancy within five years that could affect the treatment of prostate cancer or survival of the subject.
* History or current evidence of drug or alcohol abuse within the last 12 months.
* History of any illness (including psychiatric) that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the subject.
* Known hypersensitivity to any 5 alpha-reductase inhibitor or to any drug chemically related to dutasteride.

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2007-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (60):
- United States (46):
  - GSK Investigational Site, Homewood, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, San Bernardino, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Galesburg, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Jeffersonville, Indiana
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Annapolis, Maryland
  - GSK Investigational Site, Watertown, Massachusetts
  - GSK Investigational Site, Chaska, Minnesota
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Garden City, New York
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Concord, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Bala-Cynwyd, Pennsylvania
  - GSK Investigational Site, Lancaster, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Myrtle Beach, South Carolina
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Norfork, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Virginia Beach, Virginia
  - GSK Investigational Site, Williamsburg, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
- Canada (14):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Barrie, Ontario
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, North Bay, Ontario
  - GSK Investigational Site, Oakville, Ontario
  - GSK Investigational Site, Scarborough Village, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Laval, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: AVO108943 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AVO108943 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AVO108943 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AVO108943 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AVO108943 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AVO108943 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AVO108943 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Bicalutamide 50 mg/Placebo: Participants were randomly assigned to receive oral bicalutamide 50 milligrams (mg) and matching placebo once daily for 18 months. Participants who completed the 18-month treatment period with either stabilization or a positive response to their prostate cancer were offered participation in the 2-year extension phase , during which they would remain on their current treatment. A safety follow-up was conducted 16 weeks (+/-7 days) after withdrawal from investigational product (end of treatment or early withdrawal).
- Bicalutamide 50 mg/Dutasteride 3.5 mg: Participants were randomly assigned to receive oral bicalutamide 50 mg and dutasteride 3.5 mg once daily for 18 months. Participants who completed the 18-month treatment period with either stabilization or a positive response to their prostate cancer were offered participation in the 2-year extension phase, during which they would remain on their current treatment. A safety follow-up was conducted 16 weeks (+/-7 days) after withdrawal from investigational product (end of treatment or early withdrawal).
Period: Treatment Period (18 Months)
Arm/Group | Bicalutamide 50 mg/Placebo | Bicalutamide 50 mg/Dutasteride 3.5 mg
Started | 65 | 62
Completed | 27 | 31
Not Completed | 38 | 31
Not completed — Protocol-defined Stopping Criteria | 16 | 14
Not completed — Adverse Event | 7 | 6
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Physician Decision | 4 | 4
Not completed — Protocol Violation | 3 | 1
Not completed — Sponsor Terminated Study | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Non-compliance | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Period: Extension Period (24 Months)
Arm/Group | Bicalutamide 50 mg/Placebo | Bicalutamide 50 mg/Dutasteride 3.5 mg
Started | 26 (One participant who completed the Treatment Period did not participate in the Extension Period.) | 30 (One participant who completed the Treatment Period did not participate in the Extension Period.)
Completed | 11 | 7
Not Completed | 15 | 23
Not completed — Protocol-defined Stopping Criteria | 6 | 7
Not completed — Adverse Event | 3 | 4
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Physician Decision | 4 | 3
Not completed — Sponsor Terminated Study | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Non-compliance | 0 | 1
Not completed — Disease Progression | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bicalutamide 50 mg/Placebo | Bicalutamide 50 mg/Dutasteride 3.5 mg | Total
Number analyzed (Participants) | 65 | 62 | 127
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.6 (7.90) | 78.9 (5.94) | 78.3 (7.02)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 65 | 62 | 127
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 11 | 10 | 21
  American Indian or Alaska Native | 2 | 1 | 3
  Asian-Japanese Heritage | 1 | 0 | 1
  Asian-South East Asian Heritage | 0 | 1 | 1
  White-White/Caucasian/European Heritage | 51 | 50 | 101

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression
Description: Time to disease progression (PD) is defined as the interval of time between the date of the start of treatment and the date of PD. PD is defined as prostate specific antigen (PSA) progression from Baseline (PSA value is 25% and at least 2 nanograms per milliliter [ng/mL] above Baseline, confirmed by a second PSA value); PSA progression from nadir, without a 50% decrease from Baseline (PSA value is 25% and at least 2 ng/mL above nadir, confirmed by a second PSA value); PSA progression from nadir, with a 50% or more decrease from Baseline (PSA value is 50% and at least 2 ng/mL above nadir, confirmed by a second PSA value); metastatic disease (radiographic evidence of metastatic disease); death due to prostate cancer; or the receipt of post-Baseline rescue medication. PSA confirmation was not required if no subsequent PSA values were available. Participants who did not experience an event were censored at the date of the latest follow-up information.
Time Frame: Interval of time between the date of the start of treatment and the date of disease progression (up to Study Month 42)
Population: Intent-to-Treat (ITT) Population: all participants randomized to study treatment. Data were not summarized for censored participants (no disease progression).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Bicalutamide 50 mg/Placebo | Bicalutamide 50 mg/Dutasteride 3.5 mg
Number analyzed (Participants) | 41 | 40
Days | 376.9 (333.94) | 433.1 (324.25)
Statistical Analysis 1: Comparison: Bicalutamide 50 mg/Placebo vs Bicalutamide 50 mg/Dutasteride 3.5 mg; Test type: Superiority or Other; p = 0.79, Log Rank
Statistical Analysis 2: Comparison: Bicalutamide 50 mg/Placebo vs Bicalutamide 50 mg/Dutasteride 3.5 mg; Test type: Superiority or Other; Relative Risk = 0.94, 95% CI 2-sided [0.61 to 1.46] — The hazard ratio is based on the Cox proportional hazards model
Statistical Analysis 3: Comparison: Bicalutamide 50 mg/Placebo vs Bicalutamide 50 mg/Dutasteride 3.5 mg; Test type: Superiority or Other; Relative Risk Reduction = 5.62, 95% CI 2-sided [-46.14 to 39.05] — Relative Risk Reduction = 100 * (1 - Relative Risk)

2. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined as the interval of time between the date of the start of treatment and the date of treatment failure. Treatment failure is defined as PSA progression from Baseline (PSA value is 25% and at least 2 ng/mL above Baseline, confirmed by a second PSA value); metastatic disease (radiographic evidence of metastatic disease); death due to prostate cancer; or receipt of post-baseline rescue medications. PSA confirmation was not required if no subsequent PSA values were available. Participants who did not experience an event were censored at the date of the latest follow-up information.
Time Frame: Interval of time between the date of the start of treatment and the date of treatment failure (up to Study Month 42)
Population: ITT Population. Data were not summarized for censored participants (no treatment failure).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Bicalutamide 50 mg/Placebo | Bicalutamide 50 mg/Dutasteride 3.5 mg
Number analyzed (Participants) | 31 | 28
Days | 368.4 (323.94) | 457.5 (322.01)

3. Secondary Outcome: Number of Participants With PSA Response
Description: PSA response is defined as a 50% or greater decrease in PSA from Baseline, confirmed by a second PSA measurement. The time of this response was the date of the first PSA measurement that showed a 50% or greater decrease from the Baseline PSA measurement. PSA confirmation was not required if no subsequent PSA values were available.
Time Frame: Time from Baseline PSA measurement until the first PSA measurement with a 50% or greater reduction in PSA values (up to Study Month 42)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Bicalutamide 50 mg/Placebo | Bicalutamide 50 mg/Dutasteride 3.5 mg
Number analyzed (Participants) | 65 | 62
participants
  Months 1-18, n=65, 62 | 37 | 38
  Months 19-42, n=4, 7 | 0 | 0
  Overall (Months 1-42), n=65, 62 | 37 | 38

4. Secondary Outcome: Change From Baseline in Total PSA at Months 6, 12, 18, 21, and 42
Description: Change from Baseline in total PSA was measured at each scheduled post-baseline visit using a general linear model with effects for treatment and Baseline total PSA. Analysis was done using the last observation carried forward (LOCF) approach, in which missing post-Baseline values were imputed with earlier non-missing values. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Months 6, 12, 18, 21, and 42
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Median (Full Range); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Bicalutamide 50 mg/Placebo | Bicalutamide 50 mg/Dutasteride 3.5 mg
Number analyzed (Participants) | 65 | 62
Nanograms per milliliter (ng/mL)
  Month 6, n=62, 61 | -2.0 [-12.4 to 74.0] | -2.2 [-17.6 to 15.0]
  Month 12, n=62, 61 | -1.7 [-12.5 to 74.0] | -2.1 [-17.7 to 33.6]
  Month 18, n=62, 61 | -1.2 [-12.7 to 74.0] | -1.7 [-17.9 to 33.6]
  Month 21, n=26, 30 | -2.1 [-12.7 to 2.4] | -1.8 [-17.9 to 7.0]
  Month 42, n=26, 30 | -0.1 [-12.7 to 23.6] | 0.6 [-18.0 to 13.0]

5. Secondary Outcome: Number of Participants With Metastatic Disease
Description: Metastatic disease is that evidenced by a radiographic assessment. The time of metastatic disease was the date of radiographic evidence.
Time Frame: Interval of time between the date of the start of treatment and the date of radiographic evidence of metastatic disease (up to Study Month 42)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Bicalutamide 50 mg/Placebo | Bicalutamide 50 mg/Dutasteride 3.5 mg
Number analyzed (Participants) | 65 | 62
participants
  Months 1-18, n=65, 62 | 8 | 5
  Months 19-42, n=26, 30 | 1 | 1
  Overall (Months 1-42), n=65, 62 | 9 | 6

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs)/non-serious AEs were collected from the first dose of investigational product to the follow-up (FU) period (16 weeks after end of study treatment) (up to approximately Study Month 46 [42 months of treatment+16 weeks of FU]).
Description: SAEs and AEs were collected in members of the ITT Population, comprised of all participants randomized to study treatment.
Arm/Group | Bicalutamide 50 mg/Placebo | Bicalutamide 50 mg/Dutasteride 3.5 mg
Serious Adverse Events (participants affected / at risk) | 31/65 | 30/62
Other Adverse Events (participants affected / at risk) | 48/65 | 51/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bicalutamide 50 mg/Placebo (N=65) | Bicalutamide 50 mg/Dutasteride 3.5 mg (N=62)
Cerebrovascular accident (Nervous system disorders) | 2 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 0
Cellulitis (Infections and infestations) | 0 | 2
Lobar pneumonia (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Orchitis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Sepsis syndrome (Infections and infestations) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Postrenal failure (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Refractory anaemia with an excess of blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant lymphoid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bicalutamide 50 mg/Placebo (N=65) | Bicalutamide 50 mg/Dutasteride 3.5 mg (N=62)
Urinary tract infection (Infections and infestations) | 8 | 10
Oedema peripheral (General disorders) | 8 | 9
Dizziness (Nervous system disorders) | 9 | 7
Constipation (Gastrointestinal disorders) | 8 | 6
Anaemia (Blood and lymphatic system disorders) | 7 | 6
Diarrhoea (Gastrointestinal disorders) | 8 | 5
Nasopharyngitis (Infections and infestations) | 7 | 6
Fatigue (General disorders) | 7 | 5
Hot flush (Vascular disorders) | 9 | 3
Asthenia (General disorders) | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 8
Upper respiratory tract infection (Infections and infestations) | 6 | 3
Nausea (Gastrointestinal disorders) | 4 | 4
Headache (Nervous system disorders) | 6 | 2
Hypertension (Vascular disorders) | 6 | 2
Sinusitis (Infections and infestations) | 4 | 3
Urinary retention (Renal and urinary disorders) | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Vomiting (Gastrointestinal disorders) | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5
Haematuria (Renal and urinary disorders) | 6 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 4
Urinary incontinence (Renal and urinary disorders) | 4 | 2
Breast tenderness (Reproductive system and breast disorders) | 4 | 2
Ear infection (Infections and infestations) | 4 | 1
Nocturia (Renal and urinary disorders) | 5 | 0
Nipple pain (Reproductive system and breast disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.